CLINICAL TRIAL: NCT05669612
Title: Promephy - Metabolic Fate of Plant-based Proteins
Acronym: Promephy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Justin Roberts, Professor, Anglia Ruskin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R9097
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Amino Acid Change; Gastrointestinal Dysfunction
Keywords: Protein; Amino acids; Microbiota

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to each of 4 protein-related products in a double-blind, crossover, single centre study
Who Masked: Participant, Investigator
Masking Description: Protein supplements will be provided in a randomized, double-blinded manner. Both the participants and research testers will be masked from knowing the specifics of the supplement intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dairy based protein (Active Comparator): Milk protein isolate
  For bioavailability sessions: 20 grams of protein dissolved in water 200 ml water Then 50g per day (2 x 25g serves dissolved in 200 ml water) over 2 weeks
  Interventions: Dietary Supplement: Dairy based protein
- Mixed protein (Experimental): Milk and plant based protein mix
  For bioavailability sessions: 20 grams of protein dissolved in water 200 ml water Then 50g per day (2 x 25g serves dissolved in 200 ml water) over 2 weeks
  Interventions: Dietary Supplement: Mixed protein
- Plant-based protein 1 (Experimental): Plant based protein mix
  For bioavailability sessions: 20 grams of protein dissolved in water 200 ml water Then 50g per day (2 x 25g serves dissolved in 200 ml water) over 2 weeks
  Interventions: Dietary Supplement: Plant-based protein 1
- Plant-based protein 2 (Experimental): Plant based protein mix with fiber
  For bioavailability sessions: 20 grams of protein dissolved in water 200 ml water Then 50g per day (2 x 25g serves dissolved in 200 ml water) over 2 weeks
  Interventions: Dietary Supplement: Plant-based protein 2

INTERVENTIONS:
Dietary Supplement: Dairy based protein — Initial bioavailability trial, followed by 2 weeks consumption of product and follow up bioavailability trial
  Arms: Dairy based protein
Dietary Supplement: Mixed protein — Initial bioavailability trial, followed by 2 weeks consumption of product and follow up bioavailability trial
  Arms: Mixed protein
Dietary Supplement: Plant-based protein 1 — Initial bioavailability trial, followed by 2 weeks consumption of product and follow up bioavailability trial
  Arms: Plant-based protein 1
Dietary Supplement: Plant-based protein 2 — Initial bioavailability trial, followed by 2 weeks consumption of product and follow up bioavailability trial
  Arms: Plant-based protein 2

SUMMARY:
The PROMEPHY study aims to assess differences between animal versus plant-based proteins on metabolic and physiological parameters in healthy adults. It is envisaged that the results from this study will provide important and novel insights into the potential health-benefits of regular consumption of plant-based proteins. This may enable future application in products available to the consumer.

The main objective of this study is to compare the changes in serum essential amino acid bioavailability after two weeks of daily consumption of a plant-based protein mix with the changes in serum essential amino acid bioavailability after two weeks of daily consumption of a milk protein isolate. In addition this study will aim to assess the impact of different protein sources on gut microbiota and proteome composition to determine the potential health impact of consumption of plant-based proteins.

DETAILED DESCRIPTION:
Few human intervention studies have examined the short term (<4 weeks) effects of high (plant and animal) protein diets (25-30 percent of total energy intake) on intestinal microbiota composition [Beaumont et al., 2017; David et al., 2014]. One study suggests that long-term dietary patterns which involve increased consumption of protein (meat and dairy) can shift the composition of the gut microbiota towards an ecosystem in which taxa possessing proteolytic fermentation pathways are most abundant [Blachier et al., 2019]. Increased proteolytic activity is associated with increased gene expression of negative bacteria and increased uremic toxins and microbial metabolites which can potentially result in damage to the gut microstructure, activation of immune/ inflammatory responses which over a prolonged period of time may have negative health outcomes [Windey et al, 2012]. These system-level shifts in composition and metabolism hint at the complexity of metabolic interactions occurring in the host-microbiome symbiosis, but more information is needed on the processes underlying these changes.

There is current interest in the functional benefits of plant-based proteins, but with a lower bioavailability it is unclear as yet what the metabolic fate of these proteins is. Furthermore, relative to dairy proteins, plant-based sources of protein have different compounds within the structure, such as micronutrients and fibre and it is unclear if these compounds can modulate the potential negative impact of high diary protein diets on the microbiome.

The PROMEPHY study will focus on better understanding the metabolic and physiological impact of high protein diets from different (alternative) protein sources in humans. The results will provide novel insights into plant-based protein sources and may enable future application in products available to the consumer.

The primary objective of this study is to compare the changes in serum essential amino acid bioavailability after two weeks of daily consumption of a plant based protein mix with the changes in serum essential amino acid bioavailability after two weeks of daily consumption of a milk protein isolate.

Secondary objectives of this study are:

* To compare the changes in serum essential and total amino acid bioavailability after two weeks of daily consumption of a milk protein isolate, a milk and plant based protein mix, a plant based protein mix and finally a plant based protein mix with fibre.
* To compare the changes in taxonomic microbiota and proteome composition after one week and after two weeks of daily consumption of a milk protein isolate, a milk and plant based protein mix, a plant based protein mix and finally a plant based protein mix with fibre.

This is a randomised, double-blind, crossover, single centre study. It is anticipated that 15-20 healthy participants will be recruited (men and women, aged 18-50 years) for this cross-over design study (see eligibility).

Proposed methods

This study will involve participants attending an initial screening session, followed by 3 laboratory visits to the Human Physiology Laboratory at Anglia Ruskin University, Cambridge, UK, for each of 4 trials (total of 13 visits). A brief overview of the key visits are provided here:

Screening session Volunteers will initially be required to attend a study briefing session and screening assessment to confirm eligibility. This will take place at Anglia Ruskin University, Cambridge, UK. Participants will be required to provide written, informed consent and will receive information on study arrangements.Volunteers eligible for participation will be provided with stool collection material and will receive instructions on collection and storage of the stool sample. Subjects eligible for participation will then visit the Human Physiology Laboratory, Anglia Ruskin University, Cambridge, UK a further 12 times over 4 trials.This is a longitudinal, cross-over design study, with at least 6 weeks between each trial (hence the study period will last at least 32 weeks). The outline of each trial is provided below. For each trial there will be 3 visits i.e. trial 1a, 1b, 1c.

Visits 1a, 2a, 3a and 4a (same general protocol for visits 1c,2c,3c,4c) Following an overnight fast (10 hours), subjects will come to the Human Physiology Laboratory, Anglia Ruskin University, UK for a bioavailability assessment. The research team will receive a stool sample that subjects collected at home maximally three days prior to the study visit and the Bristol Stool Chart that subjects completed on the same day of the stool sample collection. Habitual dietary intake will be assessed via a mobile application (MyFitnessPal). Body weight will be measured. Subjects will consume one serving of one of the four study products (randomization at Visit 1a, one portion contains 20 grams of protein) dissolved in water 200 ml water, and consumed within 10 minutes. Blood samples will be drawn at T= -20 and -5 min (baseline) and at t= 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, and 240 min after study product intake by a qualified phlebotomist. Samples will be assessed for uremic markers (baseline only) and amino acid profiles. A gastrointestinal tolerance questionnaire will be completed at several time points (before study product intake and at 90 and 240 min). Throughout the study visits subjects are not allowed to eat, but will drink 200 ml water at T=95 and T=185 min. In addition, participants will be asked to abstain from any physical exercise other than incidental walking during the study visits. After this study visit a 2-week (± 2 days) dietary intervention will start, with the first serving at home taken in the evening. Participants will receive 50 g of protein to consume daily at home (1 x 25 g in morning and 1 x 25 g in evening), not combined with a meal. Participants will undertake a follow-up assessment 2 weeks later using the same protocol outlined above.

Visits 1b, 2b, 3b and 4b One week after visit a, participants will visit the Human Physiology Laboratory, Anglia Ruskin University, Cambridge, UK again for visit b after an overnight fast (at least 10 hours). The research team will receive a stool sample that participants collected within 3 days prior to the study visit and the Bristol Stool Chart that participants completed on the same day of the stool sample collection. Body weight will be measured. A fasting blood sample will be taken only for assessment of uremic markers.

Each trial will be separated by at least a 6 weeks washout period.

In this study four study products will be investigated:

* Product A: Milk protein isolate
* Product B: Milk and plant based Protein mix
* Product C: Plant based protein mix
* Product D: Plant based protein mix with fiber

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 50 years
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 24.9 kg/m2
3. Written informed consent
4. Willingness and ability to comply with the protocol
5. Willingness to use a method of birth control during participation in the study (women only)
6. Judged by the investigator to be in good health

Exclusion Criteria:

1. Any known ongoing medical condition that interferes significantly with absorption and digestion and/or gastrointestinal (GI) function (e.g. inflammatory bowel disease, gastroesophageal reflux disease, celiac disease, diaphragmatic hernia or diaphragmatic surgery, gastric ulcer, gastritis, gall bladder problems, pancreatitis, GI cancer, oesophageal and/or gastric surgery), in opinion of the investigator.
2. Known cardiovascular disease, disease related to the immune system and/or the respiratory system
3. Known renal or hepatic failure or known thyroid dysfunction
4. Known Diabetes Mellitus type I or type II
5. Any ongoing cancer (except for basal cell carcinoma) and/ or cancer treatment
6. Haemoglobin (Hb) in men <7.5 mmol/l and in women <7.0 mmol/l at screening
7. Any known bleeding disorder
8. Use of oral and systemic use of prokinetics, laxatives, antidiarrheals, anticoagulants within 3 weeks of Visit 1
9. Use of antibiotics within 3 months prior to Visit 1
10. Known lactose intolerance or known plant-based protein allergy
11. Adherence to a strict dietary regime (e.g. vegetarian/ vegan/ paleo/ketogenic/high protein diet or a weight loss program)
12. Use of any nutritional supplements or additional protein supplements or nutritional support within 6 weeks prior to visit 1
13. Regular heavy and/or extreme exercise (e.g. trained elite athletes) in opinion of the investigator
14. Known pregnancy and/or lactation (women only)
15. Current smoking or stopped smoking for < 1 month prior to screening (except for incidental smoking of ≤ 3 cigarettes/cigars/pipes per week on average in the last month) and willingness to stop entirely during study participation (after enrolment).
16. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women (on average during the last 6 months) or drug/ medicine abuse in opinion of the investigator
17. Participation in any other clinical study with investigational or marketed products concomitantly or within four weeks before study visit 1
18. Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the investigator
19. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Amino acid Profile | Change from beginning (day 1) to end of each trial (day 14)
  Measurement of essential amino acids (EAA; umol/L) area under the curve (iAUC) after two weeks of study product intake of plant based protein mix vs dairy protein mix

SECONDARY OUTCOMES:
Uremic blood markers | Change from beginning (day 1) to end of each trial (day 14)
  Measurement of serum uremic acids (umol/L)
Microbiota profile | Change from beginning (day 1) to end of each trial (day 14)
  Untargeted Microbiota analyses from stool samples will be performed through 16S rRNA gene sequencing using gene primers for region V3-V4
Proteome data | Change from beginning (day 1) to end of each trial (day 14)
  Proteome data from stool samples will be generated using nano-LC-LTQ-Orbitrap-MS

CONTACTS AND LOCATIONS:
Overall Officials: Justin Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blachier F, Beaumont M, Portune KJ, Steuer N, Lan A, Audebert M, Khodorova N, Andriamihaja M, Airinei G, Benamouzig R, Davila AM, Armand L, Rampelli S, Brigidi P, Tome D, Claus SP, Sanz Y. High-protein diets for weight management: Interactions with the intestinal microbiota and consequences for gut health. A position paper by the my new gut study group. Clin Nutr. 2019 Jun;38(3):1012-1022. doi: 10.1016/j.clnu.2018.09.016. Epub 2018 Sep 20. PMID 30274898
- [Background] Windey K, De Preter V, Verbeke K. Relevance of protein fermentation to gut health. Mol Nutr Food Res. 2012 Jan;56(1):184-96. doi: 10.1002/mnfr.201100542. Epub 2011 Nov 25. PMID 22121108
- [Result] Beaumont M, Portune KJ, Steuer N, Lan A, Cerrudo V, Audebert M, Dumont F, Mancano G, Khodorova N, Andriamihaja M, Airinei G, Tome D, Benamouzig R, Davila AM, Claus SP, Sanz Y, Blachier F. Quantity and source of dietary protein influence metabolite production by gut microbiota and rectal mucosa gene expression: a randomized, parallel, double-blind trial in overweight humans. Am J Clin Nutr. 2017 Oct;106(4):1005-1019. doi: 10.3945/ajcn.117.158816. Epub 2017 Sep 13. PMID 28903954
- [Result] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Result] Liu J, Klebach M, Visser M, Hofman Z. Amino Acid Availability of a Dairy and Vegetable Protein Blend Compared to Single Casein, Whey, Soy, and Pea Proteins: A Double-Blind, Cross-Over Trial. Nutrients. 2019 Nov 1;11(11):2613. doi: 10.3390/nu11112613. PMID 31683779